CLINICAL TRIAL: NCT07321808
Title: Immunogenicity, Efficacy and Safety of Recombinant Herpes Zoster Vaccine (RZV) in Frail Patients: Multicentric Prospective Study
Acronym: AID4FRAIL_RZV
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Fausto Baldanti, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AID4FRAIL_RZV
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Immunocompromised Patients
Keywords: vaccination; varicella zoster; immunogenicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Herpes zoster (HZ) is a serious health problem whose incidence and severity increase with the decline of cell-mediated immunity (CMI) because of age and immunocompromised (IC) status [4]. Subclinical reactivation are described and may boost the adaptive specific immunity. T cells play a major role in preventing reactivation of Varicella Zoster virus (VZV), with a contribution of both CD4 and CD8 T cells. Accordingly, the suppression of VZV-specific T cells preceded the occurrence of HZ. Moreover, several observations support a role of B cells in contributing to the overall protection against HZ as patients with primary antibody deficiency, common variable immunodeficiency, or patients treated with B-cell depleting therapies or Janus Kinase inhibitors (JAKis) show a higher risk of HZ. The functional effectiveness of CMI can be significantly affected by different diseases (e.g. cancer and immune-mediated inflammatory diseases, IMIDs) and/or by ongoing immune-targeted therapy, giving these patients at high risk for VZV reactivation. The new recombinant zoster vaccine (RZV) reduces the risk of HZ, and vaccination is encouraged in IC individuals, including those with cancer and IMIDs [5]. Despite the efficacy and safety of RZV in healthy adults, data on IC patients are scarce. In particular, the immunogenicity of the new vaccine in frail subjects is not fully understood. On the one hand, immunosuppressive treatments can compromise the residual immunity to VZV but also the response to RZV [6]. Several therapies are known to affect B cell response such as Rituximab or CAR T cells; other treatments reduce the T cell functionality, such as T-cell inhibitors (Cytotoxic T-lymphocyte Antigen 4-Immunoglobulin, CTLA4-Ig; abatacept), the JAKis, as well as by chemotherapy. To date, the vaccination is not approved in paediatric patients. However, the investigation of the VZV-specific immunological profile in frail paediatric patients could represent a valuable tool for understanding the potential vaccination strategies in these categories.

The study and definition of an immune profile associated with a high risk of viral in RZV vaccinated patients with IC can be useful for identifying patients' candidates for preventive antiviral treatments.

This is an observational multicentric prospective cohort study. The general objective is to assess the immunogenicity of RZV vaccination in terms of the induction of humoral and cell-mediated immune responses in selected frail (altered immunocompetence) populations, including rheumatologic, oncologic, neurologic and hematologic patients.

Primary Objective: To define the overall rate of humoral responders patients after the second dose of RZV administration.

Primary Endpoint: The rate of "humoral responders" will be defined as the percentage of patients showing ≥ 4 times of gE-specific IgG response (IU/mL) after the second dose (T1m) respect to baseline (T0) Secondary Objective 2.1: To define the overall increase of humoral response after the second dose of RZV administration.

Secondary Objective 2.2: To characterize the immunogenicity induced by RZV vaccine in the different study cohorts (rheumatologic, oncologic, neurologic and hematologic patients) Secondary Objective 2.3: To evaluate the kinetics of humoral response during the first year after the vaccination Secondary Objective 2.4: To characterize gE-specific T cell mediated response elicited by RZV vaccination in overall patients Secondary Objective 2.5: Evaluation of the incidence of adverse reactions (AR) to the RZV vaccine, local and systemic, solicited and unsolicited, within the period of four weeks after the second dose of RZV.

Secondary Objective 2.6: Evaluation of the incidence of reactivation of VZV cases after the second dose of RZV.

ELIGIBILITY:
3.1.1. Adult population (longitudinal study) General inclusion criteria Age ≥ 18 years Eligibility for RZV vaccination Written informed consent

Inclusion criteria for specific sub-groups:

Rheumatologic patients:

* rheumatoid arthritis diagnosis according to classification criteria of 1987 and/or 2018
* eligibility or in therapy with JAKis o CTLA4-Ig (monotherapy or DMARD combination)

Oncologic patients:

* confirmed histological diagnosis of solid tumour (any type)
* life expectancy ≥ 6 months
* Patients with cancer who have to start immunotherapy with or without chemotherapy/targeted therapy

Hematologic patients:

* Patients with haematological malignancy treated with drugs (chemotherapy, new drugs, target therapies) other than antibodies.
* Patients treated with anti-CD19 or CD20 or CD22 or CD30 or anti-PD1 antibodies with or without chemotherapy
* Patients receiving autologous or allogeneic transplantation or CAR-T cells

Neurologic patients:

* Multiple sclerosis (MS) diagnosis according to McDonald criteria 2017
* Eligibility or in therapy with first- or second-line immunosuppressive treatments

General Exclusion criteria No informed consent Previous HZ vaccination Documented reactions or allergies against vaccines Severe infections during the previous 3 months

3.1.2. Pediatric population (cross-sectional study) Inclusion criteria Written informed consent from parents legal tutor and child assent (depending on age) Serology for VZV positive

Hematologic patients:

* Patients with haematological malignancies treated with chemotherapy including experimental drugs and target therapies;
* Patients with haematological malignancies undergoing B-cell depleting treatments, e.g. CAR-T cell therapy or anti-CD20, antiCD22, anti-CD30, anti-CD19 monoclonal or bispecific antibodies
* Patients with haematological malignancies receiving allogeneic transplantation due to malignant or non-malignant diseases, including primary immunodeficiencies, hemoglobinopathies and acquired or inherited bone marrow failure syndrome.

Rheumatologic patients:

1. patients with connective tissue diseases (including systemic lupus erythematosus, SLE, juvenile dermathomyositis, JDM, and scleroderma) treated with B cell depleting therapies (anti-CD20);
2. patients with juvenile idiopathic arthritis (JIA) treated with TNF inhibitors. The corresponding disease control populations will be patients with the same diseases listed above, who are not receiving anti-CD20 or TNF inhibitors, respectively.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: See eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To define the overall rate of humoral responders patients after the second dose of RZV administration. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Microbiologia e Virologia, Pavia, Pavia, Italy